CLINICAL TRIAL: NCT07232992
Title: The Effectiveness of the Serratus Posterior Superior Intercostal Plane Block on Postoperative Analgesia and Recovery in Open-heart Surgery: A Prospective, Double-blind, Randomized Controlled Trial.
Brief Title: Serratus Posterior Superior Intercostal Plane Block for Postoperative Analgesia in Open-Heart Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Collaborators: Emre ULUSOY (Unknown)
Responsible Party: Principal Investigator, eralp çevikkalp, assoc prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 003
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Serratus Posterior Superior Intercostal Plane Block (SPSIPB); Open-heart Surgery
Keywords: open-heart surgery; Serratus Posterior Superior Intercostal Plane Block (SPSIPB); postoperative analgesia; parasternal block
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SPSIPB (Active Comparator): It will be administered bilaterally before the induction of general anesthesia.
  Interventions: Other: SPSIPB blcok; Other: Parasternal blocks
- Group Control (Active Comparator): Parasternal block and local infiltration at the drain insertion site.
  Interventions: Other: Parasternal blocks; Other: Local Infiltration

INTERVENTIONS:
Other: SPSIPB blcok — Under aseptic conditions, an ultrasound-guided procedure will be performed using a linear probe (GE ML6-15-D Matrix Linear). After identifying the second and third ribs, a 22-gauge, 50-mm short-bevel needle (Stimuplex Ultra®, Braun, Melsungen, Germany) will be advanced in-plane in a caudocranial direction. Following hydrodissection with 5 mL of saline to confirm correct needle placement, 20 mL of 0.25% bupivacaine will be injected bilaterally into the fascial plane.
  Arms: Group SPSIPB
Other: Parasternal blocks — Before intubation, the block will be performed under aseptic conditions using a high-frequency ultrasound probe (GE ML6-15-D Matrix Linear, Boston, USA) placed immediately lateral to the sternum after identifying the second to fourth intercostal spaces. An 50-mm echogenic block needle (Stimuplex Ultra®, Braun, Melsungen, Germany) will then be advanced using an in-plane approach from the skin toward the plane between the pectoralis major and intercostal muscles. A total of 10 mL of 0.25% bupivacaine will be injected bilaterally.
Other: Local Infiltration — Local anesthetic infiltration (10 mL of 0.25% bupivacaine) will be administered around the chest tube and mediastinal drain sites.
  Arms: Group Control

SUMMARY:
Postoperative pain following open-heart surgery is a significant challenge that may negatively affect recovery and overall clinical outcomes. Due to the risks and contraindications associated with neuraxial techniques, the use of fascial plane blocks has increased in recent years. In patients undergoing cardiac surgery, the location and intensity of postoperative pain may vary daily. However, during the first 24 hours, pain is typically most pronounced at the median sternotomy incision site and at the insertion sites of chest, mediastinal, and pleural drains.

Current postoperative analgesia practices in open-heart surgery commonly include multimodal regimens using simple analgesics such as paracetamol and nonsteroidal anti-inflammatory drugs, combined with a regional anesthesia technique such as the parasternal block. The Serratus Posterior Superior Intercostal Plane Block (SPSIPB) is an interfascial plane block that involves the injection of local anesthetic between the serratus posterior superior and intercostal muscles, providing wide dermatomal coverage from the upper cervical to lower thoracic regions. Although the technique has been used successfully in individual clinical cases, no randomized controlled studies have been conducted to evaluate its efficacy in open-heart surgery.

This study aims to compare the postoperative analgesic effectiveness of the SPSIPB with a combination of parasternal block and local anesthetic infiltration at drain insertion sites in patients undergoing open-heart surgery.

DETAILED DESCRIPTION:
Postoperative pain following open-heart surgery is a significant challenge that may negatively affect recovery and overall clinical outcomes. Due to the risks and contraindications associated with neuraxial techniques, the use of fascial plane blocks has increased in recent years. In patients undergoing cardiac surgery, the location and intensity of postoperative pain may vary daily. However, during the first 24 hours, pain is typically most pronounced at the median sternotomy incision site and at the insertion sites of chest, mediastinal, and pleural drains.

Current postoperative analgesia practices in open-heart surgery commonly include multimodal regimens using simple analgesics such as paracetamol and nonsteroidal anti-inflammatory drugs, combined with a regional anesthesia technique such as the parasternal block. The Serratus Posterior Superior Intercostal Plane Block (SPSIPB) is an interfascial plane block that involves the injection of local anesthetic between the serratus posterior superior and intercostal muscles, providing wide dermatomal coverage from the upper cervical to lower thoracic regions. Although the technique has been used successfully in individual clinical cases, no randomized controlled studies have been conducted to evaluate its efficacy in open-heart surgery.

This study aims to compare the postoperative analgesic effectiveness of the SPSIPB with a combination of parasternal block and local anesthetic infiltration at drain insertion sites in patients undergoing open-heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years with ASA physical status II-III undergoing elective open-heart surgery.

Exclusion Criteria:

Patients who do not consent to participate in the study

Patients with coagulopathy

History of allergy or toxicity to local anesthetics

Patients with hepatic or renal failure

Patients with uncontrolled diabetes mellitus

Patients with uncontrolled hypertension

Mentally disabled patients

Patients receiving chronic pain therapy (opioid use)

Use of antidepressant medication

Presence of neuropathic pain

Presence of infection at the injection site

Pregnant, suspected pregnant, or breastfeeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | 0, 2, 4, 8, 16 and 24 hours
  Fentanyl will be prepared at a concentration of 10 µg/mL, and patient-controlled analgesia (PCA) will be administered without a basal infusion, using a lock-out interval of 20 minutes and a bolus dose of 20 µg.

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | 0, 2, 4, 8, 16 and 24 hours
  Postoperative 24 hours period. Patients' pain scores will be questioned at 0, 2, 4, 8, 16 and 24 hours.
Global recovery scoring system (patient satisfaction scale)- QoR-15 | The quality of recovery will be evaluated out of a total of 150 points according to the QoR-15 test to be applied at the portoperative 24th hour.
  Researchers will use the Turkish version of the Quality Improvement Survey/QoR-15. PART A: Participants will be asked by researchers how they felt in the last 24 hours.(0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent]) 1. Able to breathe easily 2. Been able to enjoy food 3. Feeling rested 4. Have had a good sleep 5. Able to look after personal toilet and hygiene unaided 6. Able to communicate with 7. Getting support from hospital doctors and nurses 8. Able to return to work or usual home activities 9. Feeling comfortable and in control 10. Having a feeling of general well-being PART B Participants will be asked by the researchers whether they have experienced any of the following in the last 24 hours. (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor]) 11. Moderate pain 12. Severe pain 13. Nausea or vomiting 14. Feeling worried or anxious 15. Feeling sad or depressed

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Zengin EN, Yigit H, Cobas M, Salman N, Asli Demir Z. The analgesic effects of combined bilateral parasternal block and serratus anterior plane block for coronary artery bypass grafting surgery. BMC Anesthesiol. 2024 Aug 5;24(1):274. doi: 10.1186/s12871-024-02659-7. PMID 39103782